CLINICAL TRIAL: NCT01689805
Title: Do Mutations in the Filaggrin Gene Have Clinical Importance for the Treatment Outcome in Atopic Dermatitis?
Brief Title: Clinical Importance of Filaggrin Gene Mutation for Treatment Outcome in Atopic Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anita Remitz, MD, PhD, Specialist in Dermatology, Helsinki University Central Hospital
Other Study IDs: FLG-255-AR
Record Dates: First submitted 2011-06-23; First posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Filaggrin
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples are collected to investigate if the patient has a mutation in the filaggrin gene.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with atopic dermatitis
- Non-atopic controls

SUMMARY:
Atopic dermatitis is a common disease which affects about one million people in Finland at some stage of their life. In atopic dermatitis we see a superficial inflammation of the skin and a defect in skin barrier function. The filaggrin protein plays a central role in the skin barrier function and studies indicate that about 30% of patients with atopic dermatitis have a mutation in the filaggrin gene. The aim of the study is to investigate whether a mutation in the filaggrin gene affects the clinical treatment outcome in patients with atopic dermatitis. If a mutation predisposes to a worse response to treatment, this could be examined and those patients with the mutation could be given extra treatment support for their atopic dermatitis. The prevalence of filaggrin mutation in the Finnish non-atopic population is studied in the control group.

ELIGIBILITY:
Inclusion Criteria (patients with atopic dermatitis):

* Age at least 18 years
* Clinical diagnosis of atopic dermatitis
* Need for follow-up at the Skin and Allergy Hospital
* Patient gives signed informed consent to participate in this study
* Patients parents and grandparents are of Finnish origin

Inclusion Criteria (Controls):

* No history of atopy or skin disease
* Age at least 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atopic dermatitis who are followed-up at the Skin and Allergy Hospital in Helsinki for at least one year can be included in the study.
  The control population consists of non-atopic persons without any other skin disease (samples for the control population are applied for from a sample collection of the National institute for health and welfare).
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2011-06

PRIMARY OUTCOMES:
Filaggrin mutation

SECONDARY OUTCOMES:
Response to treatment | 12 months
Serum IgE | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anita Remitz, MD, PhD, Principal Investigator — Skin and Allergy Hospital, Helsinki University Central Hospital
Locations (1):
- Skin and Allergy Hospital, Departments of Dermatology and Clinical Genetics, Helsinki, Finland